CLINICAL TRIAL: NCT07192484
Title: Effects of Kinesio Taping on Gait Ability, Balance, and Neuromuscular Functions in Subacute Stroke Patients With Foot Drop
Brief Title: Effects of Kinesio Taping in Subacute Stroke Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fooyin University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KSVGH25-CT6-22
Record Dates: First submitted 2025-09-04; First posted 2025-09-25 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Stroke Gait Rehabilitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- KT group (Experimental): Receiving additional Kinesio taping
  Interventions: Behavioral: KT group
- Control group (Other): Conventional physical therapy
  Interventions: Behavioral: Conventional group

INTERVENTIONS:
Behavioral: KT group — Receiving additional KT
  Arms: KT group
Behavioral: Conventional group — Conventional physical therapy
  Arms: Control group

SUMMARY:
A study was designed to investigate the effects of KT on gait ability, balance, and neuromuscular functions in subacute stroke patients with foot drop. The study aims to evaluate the immediate and short-term effects of KT on gait ability, balance, and neuromuscular function in subacute stroke patients with foot drop. A total of 60 participants will be recruited and randomly assigned to either a control group (conventional physical therapy) or an experimental group (receiving additional KT). Both groups will receive 30 minutes of daily physical therapy. The experimental group will undergo an initial assessment before KT application, which includes (1) activation of the dorsiflexor muscles, (2) reduction of plantar flexor spasticity, and (3) stabilization of the ankle in an everted position. After taping, a second assessment will be conducted immediately, and the tape will stay applied to patient's limb for two days, followed by a third assessment. The control group will be assessed only before the intervention and after two days. Primary outcome measures include gait ability (10-meter walk test, laboratory gait parameters, and joint angles and electromyographic activity during walking). Secondary outcomes include balance (Functional reach test, Timed Up and Go test, and Activities-specific Balance Confidence Scale) and neuromuscular function assessments (muscle strength, joint range of motion, spasticity, and proprioception). This project aims to establish and validate a clinically applicable and effective KT protocol as an adjunctive gait training method for subacute stroke patients with foot drop. By enhancing independent and safe walking, this intervention may facilitate the early return to normal daily activities for stroke survivors.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20 and 80 years;
* First unilateral stroke;
* Stroke onset between at least 1 week and 1 year;
* Ability to continuously walk 10 meters with or without assistive devices;
* Presence of foot drop on the affected side during the swing phase due to insufficient ankle dorsiflexion;
* Brunnstrom stage of the affected lower limb ≥ 3;
* Presence of mild spasticity in the affected ankle plantar flexors, with a Modified Ashworth Scale score ≤ 2;
* Ability to follow simple commands

Exclusion Criteria:

* Other neurological disorders or unstable medical conditions;
* Skin allergies that interfere with the use of tape;
* Visual field defects;
* Cognitive impairment, defined as a Mini-Mental State Examination (MMSE) score < 24;
* Pusher syndrome;
* Ankle contracture;
* Hemispatial neglect;
* Poorly controlled hypertension or cardiovascular disease;
* Any other disease, apart from stroke, that may affect balance or gait.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Gait ability - 10 meter walk test | 1. Baseline (prior to KT application, Day 1) 2. Immediately after KT application (Day 1) 3. 48 hours after KT application (Day 3)
  The participant will be asked to walk at a comfortable speed along a 14-meter walkway. The examiner uses a stopwatch to record the time taken to walk the middle 10 meters, and then divides the distance (10 meters) by the time to calculate the walking speed.
Gait ability - Speed (m/s) | 1. Baseline (prior to KT application, Day 1) 2. Immediately after KT application (Day 1) 3. 48 hours after KT application (Day 3)
  The participant will be asked to walk at a comfortable speed along a 14-meter walkway. Speed (m/s) will be recorded using the commercially available portable gait analysis system (Gait Up).
Gait ability - Cadence (steps/minute) | 1. Baseline (prior to KT application, Day 1) 2. Immediately after KT application (Day 1) 3. 48 hours after KT application (Day 3)
  The participant will be asked to walk at a comfortable speed along a 14-meter walkway. Cadence (steps/minute) will be recorded using the commercially available portable gait analysis system (Gait Up).
Gait ability - Stride length (m) | 1. Baseline (prior to KT application, Day 1) 2. Immediately after KT application (Day 1) 3. 48 hours after KT application (Day 3)
  The participant will be asked to walk at a comfortable speed along a 14-meter walkway. Stride length (m) will be recorded using the commercially available portable gait analysis system (Gait Up).
Gait ability - Step length (m) | 1. Baseline (prior to KT application, Day 1) 2. Immediately after KT application (Day 1) 3. 48 hours after KT application (Day 3)
  The participant will be asked to walk at a comfortable speed along a 14-meter walkway. Step length (m) will be recorded using the commercially available portable gait analysis system (Gait Up).
Gait ability - Percentages of stance phase (%) | 1. Baseline (prior to KT application, Day 1) 2. Immediately after KT application (Day 1) 3. 48 hours after KT application (Day 3)
  The participant will be asked to walk at a comfortable speed along a 14-meter walkway. Percentages of stance phase (%) will be recorded using the commercially available portable gait analysis system (Gait Up)
Gait ability - Percentages of swing phase (%) | 1. Baseline (prior to KT application, Day 1) 2. Immediately after KT application (Day 1) 3. 48 hours after KT application (Day 3)
  The participant will be asked to walk at a comfortable speed along a 14-meter walkway. Percentages of swing phase (%) will be recorded using the commercially available portable gait analysis system (Gait Up).
Gait ability - Gait symmetry (%) | 1. Baseline (prior to KT application, Day 1) 2. Immediately after KT application (Day 1) 3. 48 hours after KT application (Day 3)
  Gait symmetry (%) will be recorded using the commercially available portable gait analysis system (Gait Up).
Gait ability - first maximum toe clearance (cm) | 1. Baseline (prior to KT application, Day 1) 2. Immediately after KT application (Day 1) 3. 48 hours after KT application (Day 3)
  The participant will be asked to walk at a comfortable speed along a 14-meter walkway. The first maximum toe clearance (cm) will be recorded using the commercially available portable gait analysis system (Gait Up).
Gait ability - second maximum toe clearance (cm) | 1. Baseline (prior to KT application, Day 1) 2. Immediately after KT application (Day 1) 3. 48 hours after KT application (Day 3)
  The participant will be asked to walk at a comfortable speed along a 14-meter walkway. The second maximum toe clearance (cm) will be recorded using the commercially available portable gait analysis system (Gait Up).
Gait ability - minimum toe clearance (cm) | 1. Baseline (prior to KT application, Day 1) 2. Immediately after KT application (Day 1) 3. 48 hours after KT application (Day 3)
  The participant will be asked to walk at a comfortable speed along a 14-meter walkway. The minimum toe clearance (cm) will be recorded using the commercially available portable gait analysis system (Gait Up).
Ankle joint range (degrees) during walking | 1. Baseline (prior to KT application, Day 1) 2. Immediately after KT application (Day 1) 3. 48 hours after KT application (Day 3)
  The participant will be asked to walk at a comfortable speed along a 14-meter walkway. Ankle joint range (degrees) during walking will be recorded using the commercially wireless system (Delsys Inc., United States).
EMG activity (µV) of tibialis anterior during walking | 1. Baseline (prior to KT application, Day 1) 2. Immediately after KT application (Day 1) 3. 48 hours after KT application (Day 3)
  The participant will be asked to walk at a comfortable speed along a 14-meter walkway. EMG activity (µV) of tibialis anterior during walking will be recorded using the commercially wireless system (Delsys Inc., United States).
EMG activity (µV) of gastrocnemius during walking | 1. Baseline (prior to KT application, Day 1) 2. Immediately after KT application (Day 1) 3. 48 hours after KT application (Day 3)
  The participant will be asked to walk at a comfortable speed along a 14-meter walkway. EMG activity (µV) of gastrocnemius during walking will be recorded using the commercially wireless system (Delsys Inc., United States).

SECONDARY OUTCOMES:
Functional reach test | 1. Baseline (prior to KT application, Day 1) 2. Immediately after KT application (Day 1) 3. 48 hours after KT application (Day 3)
  Participant is asked to stand by the wall without leaning against it, with hands clenched into fists and arms raised forward to shoulder height with the shoulder joints flexed at 90 degrees. The examiner records the position of the participant's third metacarpal bone as the starting point. Then, while keeping both arms raised, the participant is instructed to lean the body forward as far as possible. The examiner records the farthest position of the third metacarpal bone as the endpoint. The test result is determined by subtracting the starting point from the endpoint.
Timed Up and Go test | 1. Baseline (prior to KT application, Day 1) 2. Immediately after KT application (Day 1) 3. 48 hours after KT application (Day 3)
  In this test, a distance of three meters is marked on the floor, with a chair equipped with armrests and a backrest placed at one end. The participant is first asked to sit on the chair with their back against the backrest. When the examiner gives the start signal, the participant is required to rise from the chair, walk forward three meters at their usual walking speed to the marked line, turn around, walk back, and sit down on the chair again. The time taken from the moment the examiner gives the start signal until the participant has seated themselves back on the chair is recorded using a stopwatch.
Activities-specific Balance Confidence Scale | 1. Baseline (prior to KT application, Day 1) 2. Immediately after KT application (Day 1) 3. 48 hours after KT application (Day 3)
  This scale is a questionnaire designed to assess the participant's self-confidence in maintaining balance and avoiding falls in 16 situations that may be encountered in the community. Each of the 16 items is scored starting from 0, where 0 indicates no confidence at all. Scores are given in increments of 10, up to a maximum of 100, with 100 representing complete confidence.
Muscle strength | 1. Baseline (prior to KT application, Day 1) 2. Immediately after KT application (Day 1) 3. 48 hours after KT application (Day 3)
  Muscle strength of the ankle dorsiflexors will be measured using a handheld dynamometer (MicroFET3; Hoggan Health Industries, Salt Lake City, UT, USA). The participant lies supine on a treatment table with both feet hanging over the edge. The dynamometer is positioned on the dorsal aspect of the metatarsophalangeal joints to assess dorsiflexor strength. During the test, the examiner holds the dynamometer stationary while the participant exerts maximal force against it. Each contraction is sustained for 5 seconds, repeated three times, with a 10-second rest interval between trials. The mean value of the peak force obtained across the three trials will be used for analysis.
Joint range of motion | 1. Baseline (prior to KT application, Day 1) 2. Immediately after KT application (Day 1) 3. 48 hours after KT application (Day 3)
  Active range of motion (ROM) of ankle dorsiflexion and plantarflexion will be measured using a goniometer. The participant is positioned in a high sitting posture. The fulcrum of the goniometer is placed over the lateral malleolus of the ankle, with the stationary arm aligned parallel to the lateral aspect of the fibula and the moving arm aligned parallel to the fifth metatarsal. Starting from the neutral position at 0°, the participant is instructed to perform maximal active dorsiflexion followed by plantarflexion.
Spasticity | 1. Baseline (prior to KT application, Day 1) 2. Immediately after KT application (Day 1) 3. 48 hours after KT application (Day 3)
  The degree of ankle muscle spasticity will be assessed using the Modified Ashworth Scale (MAS). During the test, the joint is passively moved through its range of motion with a quick stretch to determine the presence of resistance. The scale consists of six grades (0, 1, 1+, 2, 3, 4), where a score of 0 indicates normal muscle tone and higher scores represent increasing severity of spasticity.
Proprioception | 1. Baseline (prior to KT application, Day 1) 2. Immediately after KT application (Day 1) 3. 48 hours after KT application (Day 3)
  Proprioception will be assessed using the inclinometer function of the muscle strength and angle measurement device (MicroFET3; Hoggan Health Industries, Salt Lake City, UT, USA) on the affected foot. The participant is seated on a treatment table with eyes closed and the knee extended, with the ankle positioned at 0° dorsiflexion as the starting position. The inclinometer is placed on the dorsum of the foot. The examiner passively positions the ankle to a target dorsiflexion or plantarflexion angle, and the participant is instructed to maintain this position for 10 seconds before returning to the starting position. The participant is then asked to actively reproduce the target angle. Both the examiner-set angle and the participant-reproduced angle are recorded, and the error between the two values is used to represent proprioceptive acuity.

IPD SHARING:
Plan to Share IPD: No